CLINICAL TRIAL: NCT01395251
Title: Phase II/III Study of Oral Prednisolone Test in Patients With Rheumatoid Arthritis
Brief Title: Diagnostic Value of Oral Prednisolone Test for Rheumatoid Arthritis
Acronym: TryCort
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rheumazentrum Ruhrgebiet (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Jürgen Braun, Professor of Rheuamtology, Rheumazentrum Ruhrgebiet
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: TryCort
Record Dates: First submitted 2011-07-12; First posted 2011-07-15 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; diagnosis; sensitivity; glucocorticoids
MeSH Terms: conditions — Arthritis, Rheumatoid; Disease; Hypersensitivity | interventions — Prednisolone; Glucocorticoids

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prednisolone (Other): Patients with suspicious of rheumatoid arthritis will undergo a prednisolone test with 20 mg per day for 3 days after 2 days of therapy with paracetamol 500 mg twice for 2 days.
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Prednisolone — prednisolone 20 mg once a day per os for 3 subsequent days
  Other Names: glucocorticoids

SUMMARY:
Rheumatoid arthritis is an inflammatory joint disease often leading to progressive joint destruction. To prevent disability caused by inflamed joints early diagnosis is important. Early diagnosis might be a challenge because the diagnosis is mostly based on clinical signs like swelling of small joints. In clinical practice a therapy with prednisolone is started although the patients do not have an exact diagnosis. In this cases the prednisolone might serve as a diagnostic test for an inflammatory process.

The objective of this study is to investigate the diagnostic value of oral prednisolone test for rheumatoid arthritis.

DETAILED DESCRIPTION:
Rheumatoid arthritis is with a prevalence of 2% an important inflammatory joint disease which often leads to impaired functioning and reduced quality of life. Early diagnosis is an important step forward to prevent progressive joint destruction. The classification criteria for rheumatoid arthritis published in 2010 are based on clinical signs (such as swelling) and laboratory findings (such as rheumatoid factor) (Aletaha D 2010). Because its diagnosis is based on clinical signs the early diagnosis for rheumatoid arthritis might be a challenge in daily clinical care.

In clinical practice a therapy with prednisolone is started although the patients do not have an exact diagnosis. It has been shown that the start of early low-dose prednisolone decreases the rate of joint destruction after two years of therapy (Kirwan JR 1995, Wassenberg S 2005). Thus, prednisolone might have effects comparable to that of disease-modifying antirheumatic drugs.

The objective of this study is to investigate the diagnostic value of oral prednisolone test for rheumatoid arthritis. The hypothesis is that in patients with rheumatoid arthritis the prednisolone test will be positive in 80% of the patients whereas positive in just 20% of patients with osteoarthritis of the hand. Positive prednisolone test is defined as a 30% improvement of the symptoms in finger and wrist on a numeric rating scale from 0-100.

Patients with suspicious of rheumatoid arthritis will undergo a prednisolone test with 20 mg per day for 3 days after 2 days of therapy with paracetamol 500 mg twice. After this period the patients will be asked to rate their benefit in improving pain and reducing swelling of wrist and finger joints on a numeric rating scale (0-100 % improvement in steps of 20%). A positive response In addition, demographics and clinical parameter including the compound measure for disease activity DAS-28 will be collected. A patient with a positive prednisolone test will receive standard care for rheumatoid arthritis onward. Patients with a negative prednisolone test will receive standard care for hand and finger osteoarthritis onward. At week 12 all patients will be seen again to reassess the former diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* pain in wrist and fingers without known diagnosis since more than 6 weeks, minimum of pain on a numerical rating scale 4 (out of 10)

Exclusion Criteria:

* rheumatoid arthritis
* psoriatic arthritis
* psoriasis vulgaris
* vasculitis
* gouty arthritis
* Current glucocorticoidmedication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-02; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Rate of true diagnosis of rheumatoid arthritis after positive prednisolone test | 3 months
  Positive prednisolone test: change of more than 40% (on a NRS 0-100%) in painful joints after 3 days of therapy with prednisolone 20 mg/d
Rate of true negative diagnosis of rheumatoid arthritis after positive prednisolone test | 3 months
  Positive prednisolone test: change of more than 40% (on a NRS 0-100%) in painful joints after 3 days of therapy with prednisolone 20 mg/d
Negative predictive value | 3 months
Positive predictive value | 3 months

SECONDARY OUTCOMES:
clinical characteristics of patients with early RA | 3 months
change of disease activity | 3 months
  assessed with DAS-28
change of functioning | 3 months
  assessed with HAQ

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Braun, MD, Principal Investigator — Rheumazentrum Ruhrgebiet, Herne, Germany
Locations (1):
- Rheumazentrum Ruhrgebiet, Herne, Germany

REFERENCES:
- [Background] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum. 2010 Sep;62(9):2569-81. doi: 10.1002/art.27584. PMID 20872595
- [Background] Wassenberg S, Rau R, Steinfeld P, Zeidler H. Very low-dose prednisolone in early rheumatoid arthritis retards radiographic progression over two years: a multicenter, double-blind, placebo-controlled trial. Arthritis Rheum. 2005 Nov;52(11):3371-80. doi: 10.1002/art.21421. PMID 16255011
- [Background] Kirwan JR. The effect of glucocorticoids on joint destruction in rheumatoid arthritis. The Arthritis and Rheumatism Council Low-Dose Glucocorticoid Study Group. N Engl J Med. 1995 Jul 20;333(3):142-6. doi: 10.1056/NEJM199507203330302. PMID 7791815
- [Derived] Kiltz U, von Zabern C, Baraliakos X, Heldmann F, Mintrop B, Sarholz M, Krause D, Dybowski F, Kalthoff L, Braun J. Diagnostic value of a 3-day course of prednisolone in patients with possible rheumatoid arthritis - the TryCort study. Arthritis Res Ther. 2017 Apr 7;19(1):73. doi: 10.1186/s13075-017-1279-z. PMID 28388956